CLINICAL TRIAL: NCT00669149
Title: Anticoagulant Treatments Evaluation During Percutaneous Coronary Angioplasty in Stable Patients
Brief Title: Anticoagulant Treatments and Percutaneous Coronary Angioplasty
Acronym: TACA
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: recruitment difficulties
Sponsor: Centre Hospitalier de PAU (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHPAU 2007/01
Record Dates: First submitted 2008-04-25; First posted 2008-04-29 (Estimated); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Coronary Artery Disease
Keywords: ptca; antiaggregant therapy; anticoagulant therapy
MeSH Terms: conditions — Coronary Artery Disease | interventions — Clopidogrel; Aspirin; Heparin; Enoxaparin; bivalirudin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): group without anticoagulant therapy
  Interventions: Drug: clopidogrel + aspirin
- 2 (Active Comparator): group with heparin
  Interventions: Drug: heparin + clopidogrel + aspirin
- 3 (Active Comparator): group with enoxaparin
  Interventions: Drug: enoxaparin + clopidogrel + aspirin
- 4 (Active Comparator): group with bivalirudin
  Interventions: Drug: bivalirudin + clopidogrel + aspirin

INTERVENTIONS:
Drug: clopidogrel + aspirin
  Other Names: Plavix Kardégic
  Arms: 1
Drug: heparin + clopidogrel + aspirin
  Other Names: héparine Choay Plavix Kardégic
  Arms: 2
Drug: enoxaparin + clopidogrel + aspirin
  Other Names: Lovenox Plavix Kardégic
  Arms: 3
Drug: bivalirudin + clopidogrel + aspirin
  Other Names: Angiox Plavix Kardégic
  Arms: 4

SUMMARY:
The purpose of this study is to determine whether adjunction of intravenous anticoagulant therapy (enoxaparin, HNF, bivalirudin) to antiaggregation with clopidogrel and aspirin improves in-hospital results of percutaneous transluminal coronary angioplasty (ptca) in selected patients.

DETAILED DESCRIPTION:
* Background : We don't know if using IV anticoagulant therapy is necessary for percutaneous coronary angioplasty in stable patients.
* Purpose : to compare efficacy and security of use or not of different anticoagulant treatments during percutaneous coronary angioplasty in patients with double antiaggregant therapy.
* Abstract : In stable patients pretreated with double antiaggregant therapy use of IV anticoagulants has not been yet evaluated during angioplasty. In this prospective randomized trial we want to compare in such patients the efficacy and security of the administration of IV heparin, IV enoxaparin, IV bivalirudin and no use of anticoagulant during coronary angioplasty. We will evaluate in each group ischaemic events (clinic, ECG and biology) and haemorrhagic events (clinic, biology) with a one month follow up.
* Primary outcome: ischaemic events via troponin Ic measurements during 24 hours post procedure.
* Secondary outcomes: haemorrhagic events : clinical and biological evaluation (Hb, Ht, TIMI score)
* Study design : monocentric randomized clinical trial type therapeutic equivalence phase IV.
* Interventions : In patients prepared with therapeutic association (aspirin clopidogrel) comparison between use or no of anticoagulant (IV heparin, IV enoxaparin or IV bivalirudin).
* Number of subjects : 120 per group (total of 480).
* Statistical analysis : multivariate analysis with logistic regression models : each end point (troponin Ic increase, haemoglobin decrease, …) will be explicated with treatment group and other covariates (sex, age, creatinine, …).

ELIGIBILITY:
Inclusion Criteria:

* stable angina pectoris or silent ischaemia

Exclusion Criteria:

* instable angina or ACS (Acute Coronary Syndrome)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2008-06; Primary Completion 2013-08-03 (Actual); Study Completion 2013-08-03 (Actual)

PRIMARY OUTCOMES:
ischaemic events via troponin Ic measurements during 24 hours post procedure | 24 hours

SECONDARY OUTCOMES:
haemorrhagic events : clinical and biological evaluation | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas DELARCHE, MD, Principal Investigator — CH de Pau
Locations (1):
- Centre Hospitalier de Pau, Pau, Pyrénées-Atlantiques, France